CLINICAL TRIAL: NCT04483076
Title: A Prospective, Multicenter, Randomized, Controlled Phase III Study Evaluating Different Cycles of Oxaliplatin Combined With S-1 (SOX) as Neoadjuvant Chemotherapy for Patients With Locally Advanced Gastric Cancer: RESONANCE-II Trial
Brief Title: Oxaliplatin Combined With S-1(SOX) Neoadjuvant Chemotherapy for Different Cycles in Patients With Gastric Cancer
Acronym: RESONANCE-II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Prof., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESONANCE-II
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer; Chemotherapy Effect
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients will be pre-enrolled and receive three cycles of SOX. After randomization, patients in Arm A will receive three more cycles of SOX (six cycles of neoadjuvant chemotherapy with SOX in total) followed by D2 gastrectomy.
  Interventions: Drug: Chemotherapy drug; Procedure: Gastrectomy; Procedure: Laparoscopic exploration
- Arm B (Active Comparator): Patients will be pre-enrolled and receive three cycles of SOX. After randomization, patients in Arm B will receive D2 gastrectomy (three cycles of neoadjuvant chemotherapy with SOX in total).
  Interventions: Drug: Chemotherapy drug; Procedure: Gastrectomy; Procedure: Laparoscopic exploration

INTERVENTIONS:
Drug: Chemotherapy drug — The preoperative SOX chemotherapy consists of three-week cycles of intravenously administered oxaliplatin 130 mg/m2 on day 1 and orally administered S-1 40-60 mg twice a day (BID) on day 1 to 14. The dose of S-1 depends on body surface area (BSA): 40mg BID for BSA < 1.25 m2; 50mg BID for 1.25 m2 < BSA <1.5 m2; 60mg BID for BSA > 1.5 m2. Day 15 to day 21 is the rest period.
Procedure: Gastrectomy — Surgery is planned 3-4 weeks after the last cycle of chemotherapy. A standard D2 radical laparoscopic gastrectomy is recommended. The extent of gastric resection and lymphadenectomy were performed as per the treatment guidelines. Reconstruction after gastrectomy was decided by the surgeon. All operations are performed by well trained and experienced surgical team to guarantee the quality of surgery, including harvesting more than 16 lymph nodes.
Procedure: Laparoscopic exploration — Laparoscopic exploration is to detect occult peritoneal metastases and inspect the primary lesion, liver, diaphragm, pelvic organs, bowel and omentum according to the standard acquirements reported before. Patients with any patterns of distant metastases, suggestive of distant metastasis (M1), will be excluded from the trial.

SUMMARY:
RESONANCE-II trial is a prospective, multicenter, randomized, controlled phase III study which will enroll 524 patients in total. Patients with eligibility will be registered, pre-enrolled and receive three cycles of SOX. Then, tumor response evaluation will be carried out. Those who achieve stable disease or progressive disease will be excluded. Patients achieving complete response or partial response will be enrolled and assigned into either group A for another three cycles of SOX (six cycles in total) followed by D2 surgery and group B for D2 surgery (three cycles in total). The primary endpoint is the rate of pathological complete response and the secondary endpoints are R0 resection rate, three-year disease-free survival, five-year overall survival and safety.

DETAILED DESCRIPTION:
RESONANCE-II trial is a prospective, multicenter, randomized, controlled phase III study which was designed to evaluate the efficacy and safety of different cycles of SOX as neoadjuvant chemotherapy for patients with locally advanced gastric cancer. All patients with eligibility will be registered, pre-enrolled and receive three cycles of SOX. Then, tumor response evaluation will be carried out according to the Response Evaluation Criteria for Solid Tumors (RECIST) 1.1. Those who achieve stable disease (SD) or progressive disease (PD)will be excluded. Patients achieving complete response (CR) or partial response (PR) will be enrolled and assigned into either group A (six cycles of neoadjuvant chemotherapy with SOX) for another three cycles of SOX followed by D2 surgery and group B (three cycles of neoadjuvant chemotherapy with SOX) for D2 surgery. The primary endpoint is the rate of pathological complete response (pCR%) and the secondary endpoints are R0 resection rate, three-year disease-free survival (3-y DFS), five-year overall survival (5-y OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Non-bedridden, aged 18 to 70 years old;
2. Eastern Cooperative Oncology Group (ECOG) score is 0 to 1;
3. Histologically confirmed gastric adenocarcinoma;
4. Stage III (American Joint Committee on Cancer (AJCC) TNM staging system 8th edition) gastric cancer confirmed by enhanced computer tomography (enhanced CT) and laparoscopic exploration (endoscopic ultrasonography (EUS) and magnetic resonance imaging (MRI) if necessary);
5. The research center and the surgeon have the ability to complete standard D2 radical gastrectomy, and the gastrectomy can be tolerated by the patient;
6. Laboratory test criteria: peripheral blood hemoglobin (Hb) ≥ 90 g/L, neutrophil absolute count ≥ 3×109 /L, platelet count (PLT) ≥ 100×109 /L, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal (ULN), total bilirubin ≤ 1.5×ULN, serum creatinine (SCr) ≤ 1.5×ULN, and serum albumin (ALB) ≥ 30 g/L;
7. Patients with heart disease, the echocardiogram showed that the left ventricular ejection fraction ≥ 50%, the electrocardiogram (ECG) is basically normal within 4 weeks before operation and without no obvious symptoms are acceptable;
8. There is no serious underlying disease that could lead to an expected life expectancy < 5 years;
9. Willing to sign the inform consent for participation and publication of results.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Positive pregnancy test for women in childbearing age. Menopausal women without menstruation for at least 12 months can be regarded as women with no possibility of getting pregnant;
3. Refuse to birth control during the study;
4. Received any chemotherapy, radiotherapy or immunotherapy before;
5. History of other malignant diseases in the last five years (except for cervical carcinoma in situ);
6. History of uncontrolled central nervous system diseases, which could influence the compliance;
7. History of severe liver diseases, renal diseases or respiratory diseases; Uncontrolled diabetes and hypertension; Clinically severe heart disease, such as congestive heart failure, symptomatic coronary heart disease, uncontrolled arrhythmia, or a history of myocardial infarction in the last six months;
8. History of dysphagia, complete or partial gastrointestinal obstruction, active gastrointestinal bleeding and gastrointestinal perforation;
9. On steroid treatment after organ transplant;
10. With uncontrolled severe infections;
11. Known dihydropyrimidine dehydrogenase deficiency (DPD);
12. Anaphylaxis to any research drug ingredient;
13. Known peripheral neuropathy (> NCI-CTC AE 1). Patients with only disappearance of deep tendon reflex need not to be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Postoperative, 2 years
  The pCR rate is defined as the rate of patients achieving pCR.

SECONDARY OUTCOMES:
R0 resection rate | Postoperative, 2 years
  The R0 resection rate is defined as the rate of R0 resection.
Three-year disease-free survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 70 months
  The DFS is defined as the period from the time of surgery to recurrence or death.
Five-year overall survival | From date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 90 months
  The OS is defined as the period from the time of surgery to death or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China